CLINICAL TRIAL: NCT03846817
Title: Optimization of the Diagnostic Process and Physiotherapist-led Treatment of Patients With Femoroacetabular Impingement Syndrome: a Prospective Cohort Study
Brief Title: Diagnosis and Treatment of Patients With Femoroacetabular Impingement Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: La Trobe University (Other); Duke University (Other)
Responsible Party: Principal Investigator, Lasse Ishøi, Principal Investigator, Hvidovre University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Physio treatment FAI
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Participants will be blinded to the potential value of the diagnostic findings, such as response to intra-articular hip injection.
  Outcome assessor will be blinded to diagnostic findings, such as response to intra-articular hip injection.
  Care Provider (Physiotherapist supervising the intervention) will be blinded to diagnostic findings, such as response to intra-articular hip injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAIS with intra-articular hip pain (Experimental): 12-week of semi-standardized, progressive physiotherapist-led treatment supervised by a physiotherapist blinded to clinical and objective findings.
  The treatment program will consist of one weekly exercise training session at Hvidovre Hospital supervised by a physiotherapist and twice-weekly unsupervised exercise training sessions performed at home for a consecutive period of 12-weeks (12 supervised sessions; 24 unsupervised sessions).
  In conjunction with the physiotherapist-led treatment, participants will be advised to modify potential aggravating physical activitie, and gradually increase their level of activity during the treatment period.
  Interventions: Other: Physiotherapist-led treatment
- FAIS without intra-articular hip pain (Experimental): 12-week of semi-standardized, progressive physiotherapist-led treatment supervised by a physiotherapist blinded to clinical and objective findings.
  The treatment program will consist of one weekly exercise training session at Hvidovre Hospital supervised by a physiotherapist and twice-weekly unsupervised exercise training sessions performed at home for a consecutive period of 12-weeks (12 supervised sessions; 24 unsupervised sessions).
  In conjunction with the physiotherapist-led treatment, participants will be advised to modify potential aggravating physical activitie, and gradually increase their level of activity during the treatment period.
  Interventions: Other: Physiotherapist-led treatment

INTERVENTIONS:
Other: Physiotherapist-led treatment — 12-week of semi-standardized, progressive physiotherapist-led treatment aiming to increase hip muscle strength and load capacity.
  Other Names: Exercise-based treatment

SUMMARY:
This prospective study with a two-group comparison design investigates the effectiveness of 12-weeks of semi-structured and supervised physiotherapist-led treatment on self-reported hip and groin function in patients with femoroacetabular impingement syndrome with and without intra-articular hip pain. Determination of intra-articular hip pain is based on pain relief following an ultrasound-guided intra-articular anesthetic hip injection performed prior to commencing treatment.

DETAILED DESCRIPTION:
The treatment of femoroacetabular impingement syndrome (FAIS) consists of wait-and-see, physiotherapist-led treatment, and/or hip surgery. The primary indication for hip surgery is based on imaging findings, however, limited correlation has been observed between such findings and hip symptoms. As patients with FAIS often show physical impariments, such as impaired hip muscle function, physiotherapist-led treatment aiming to address such factors may be effective in improving hip function and pain in some patients. However, several factors may confound the effect of physiotherapist-led treatement of FAIS, such as whether the patient presents with intra-articular hip joint pain or not.

Thus, the purpose of this prospective study with a two-group comparison design is to investigate the effect of 12-weeks of physiotherapist-led treatment on self-reported hip and groin function, measured with the Copenhagen Hip and Groin Outcome Score (HAGOS), in subjects diagnosed with FAIS, but with and without intra-articular hip pain. Determination of intra-articular hip pain is based on the response to an ultrasound-guided intra-articular anesthetic hip injection performed prior to commencing treatment.

Subjects diagnosed with FAIS based on symptoms, clinical signs and imaging findings will be prospectively recruited from a specialized outpatient hip and groin clinic at Hvidovre Hospital. Following inclusion subjects undergo 12-weeks of semi-structured and supervised physiotherapist-led treatment. The primary outcome measure is the between-group (intra-articular pain vs. no intra-articular pain) difference in mean change of the HAGOS sport subscale from baseline (week 0) to follow-up (week 12).

The primary outcome measure will be publised in the primary paper, which will also include information on between-group difference in change in hip muscle strength and single-leg hop performance as secondary outcome measures.

Secondary papers will be reported with a clear reference to the primary paper.

The sample size calculation is based on the primary outcome measure, being the between-group (intra-articular pain vs. no intra-articular pain) difference in change in the HAGOS Sport subscale following 12 weeks of physiotherapist-led treatment. Based on an expected 1/1 recruitment ratio between subjects with and without intra-articular hip pain and a clinically relevant between-group contrast in change of 15 points corresponding to a moderate effect size 0.6 (Cohen's d), a power and alpha value of 80% and 0.05, respectively, 44 subjects in each group is adequate (G*power software, v.3.1, Heinrich-Heine-Universität, Düsseldorf, Germany). To minimize the risk of underpowering the study in case of uneven allocation to groups, based on the intra-articular anesthetic hip injection, inclusion of participants will continue until a minimum of 55 (44 including 25% dropouts in each group) subjects has been recruited in each group. A blinded member of the research team will be responsible for monitoring this.

ELIGIBILITY:
Inclusion Criteria:

* Activity-related longstanding hip and/or groin pain for >3 months
* Known anterior and/or medial groin pain during the FADIR test with a pain severity of ≥2/10 on NRS.
* Radiological findings on plain radiographs of cam morphology defined as alpha angle >55° on a lateral view.

Exclusion Criteria:

* Inguinal-related groin pain diagnosed according to Doha Agreement.
* Pubic-related groin pain diagnosed according to Doha Agreement.
* Evidence of pre-existing hip osteoarthritis, defined as a joint space width <3 mm at the lateral sourcil on anterior-posterior pelvic radiograph.
* Previous hip pathology such as Perthes' disease, slipped upper femoral epiphysis, hip dysplasia defined as a Lateral Center Edge Angle <25°, or avascular necrosis.
* Other causes of hip and groin pain identified by the orthopedic surgeon during the clinical examination, such as stress fracture of the femoral neck, referred pain from the facet joint, referred pain from the sacroiliac joint, or other competing diagnosis (rheumatoid arthritis, cancer etc.)
* Previous hip injury such as acetabular fracture, hip dislocation, or femoral neck fracture.
* Previous intra- or extra-articular hip surgery.
* Pregnant.
* Intra-articular steroid hip injection during the preceding 3 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-03-12 (Estimated); Study Completion 2021-03-12 (Estimated)

PRIMARY OUTCOMES:
Change in HAGOS Sport subscale | 12 weeks
  The primary outcome measure is the between-group (intra-articular pain vs. no intra-articular pain) difference in change in self-reported hip and groin function, measured with the Copenhagen Hip and Groin Outcome Score (HAGOS) Sport subscale from baseline to follow-up in subjects diagnosed with FAIS.
  The HAGOS Sport subcale is scored on a scale from 0 (extreme hip and groin problems) to 100 (no hip and groin problems).

SECONDARY OUTCOMES:
Change in HAGOS subscales | 12 weeks
  Between-group (intra-articular pain vs. no intra-articular pain) difference in change in self-reported hip and groin function, measured with the Copenhagen Hip and Groin Outcome Score (HAGOS; all subscales exept Sport) from baseline to follow-up in subjects diagnosed with FAIS.
  The HAGOS subcales are scored on a scale from 0 (extreme hip and groin problems) to 100 (no hip and groin problems).
Change in hip peak torque | 12 weeks
  Between-group (intra-articular pain vs. no intra-articular pain) difference in change in peak isometric hip torque (Nm/kg) of abduction, adduction, extension, and flexion.
Change in hip rate of torque development | 12 weeks
  Between-group (intra-articular pain vs. no intra-articular pain) difference in change in 0-100 ms and 0-200 ms rate of torque development (Nm/s/kg) of abduction, adduction, extension, and flexion
Change in single leg hop performance | 12 weeks
  Between-group (intra-articular pain vs. no intra-articular pain) difference in change in reactive strength index obtained during a single leg drop jump test
Change in isometric adduction squeeze torque | 12 weeks
  Between-group (intra-articular pain vs. no intra-articular pain) difference in change in peak isometric hip adduction squeeze torque (Nm/kg)
Return to sport | 12 weeks
  Obtained at follow-up (week 12) using a return to sport questionnaire to determine the proportion the patients who have returned to preinjury sport at preinjury level including optimal sport performance in each group (intra-articular pain vs. no intra-articular pain).
  The outcome will be reported as proportion/frequency.
Treatment expectations and fulfilment of expectations | 12 weeks
  Treatment expectations and fulfilment of expectations will be obtained using a modified version of a questionnaire previously used and validated for patients undergoing spine surgery, which has been used previously to assess treatment expectations and fulfilment of treatment expectations in patients undergoing surgery for FAIS. Expectations and fulfilment are assessed on a 5-point Likert scale as: much better (0), better (1), somewhat better (2), unchanged (3), worse (4).
Patient acceptable symptom state | 12 weeks
  Patient Acceptable Symptom State (PASS) will be assessed at 12-weeks follow-up. The PASS defines a level of symptoms that discriminates between feeling well and unwell. Subjects will be instructed to answer the following question with yes/no: ''Taking into account all the activities you have during your daily life, your level of pain, and also your functional impairment, do you consider that your current state is satisfactory?''
  The outcome will be reported as proportion/frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Ishøi, Principal Investigator — Sports Orthopedic Research Center - Copenhagen (SORC-C), Hvidovre Hospital; Per Hölmich, Study Director — Sports Orthopedic Research Center - Copenhagen (SORC-C), Hvidovre Hospital; Kristian Thorborg, Study Director — Sports Orthopedic Research Center - Copenhagen (SORC-C), Hvidovre Hospital; Joanne Kemp, Study Chair — La Trobe Sport and Exercise Medicine Research Centre, La Trobe University; Michael Reiman, Study Chair — Duke University Medical Center, Duke University
Locations (1):
- All part of the study is conducted at Department of Orthopedic Department, Hvidovre Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided